CLINICAL TRIAL: NCT01300195
Title: Factors Predicting Persistent Post-surgical Pain After Video-assisted Thoracic Surgery (VATS)
Brief Title: Prediction of Persistent Postsurgical Pain After Video-assisted Thoracic Surgery (VATS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Dept. of thoracic Surgery (Ambiguous); Dept. of cardio-thoracic anaesthesia (Ambiguous); Dept. Surgical PAthophysiology (Ambiguous); all Blegdamsvej 9, 2100-Copenhagen, Denmark (Unknown)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H4-2010-118#0
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Pain, Postoperative
Keywords: VATS; standardized surgery; persistent pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood used to detect genetic polymorphism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer surgery: Patients undergoing video-assisted thoracic surgery

SUMMARY:
Prospective cohort study of factors predisposing to persistent post surgical pain after video-assisted thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Elective lung cancer surgery (VATS)

Exclusion Criteria:

* do not understand Danish
* cognitive reduction
* bilateral procedure planned
* previous thoracic surgery
* pregnant or nursing
* known nerve affection from other cause
* alcohol/substance abuse
* inability to cooperate to pain scoring/sensory examination
* > 5 mg methylprednisolone/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-11 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Persistent post surgical pain | 3 months
  Pain intensity (Numerical Rating Scale)
Analgesic use | 3 months
  type(s) and amount of analgesics used

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark

REFERENCES:
- [Derived] Werner MU, Ringsted TK, Kehlet H, Wildgaard K. Sensory testing in patients with postthoracotomy pain syndrome: Part 1: mirror-image sensory dysfunction. Clin J Pain. 2013 Sep;29(9):775-83. doi: 10.1097/AJP.0b013e318277b646. PMID 23328340